CLINICAL TRIAL: NCT01299142
Title: Phase I Study of Human Monoclonal Antibody (FGI-101-1A6) in Normal Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Study of Human Monoclonal Antibody (FGI-101-1A6)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Functional Genetics Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Michael Goldblatt, CEO, Functional Genetics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FGI-101-CP002; W911NF-11-C-0029 (Other Grant/Funding Number: W911NF-11-C-0029)
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Influenza
Keywords: Influenza; antibodies; monoclonal; virus
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FGI-101-1A6 (Experimental): Intervention: Drug-FGI-101-1A6
  Interventions: Drug: FGI-101-1A6
- Placebo (Placebo Comparator): Intervention: Drug-Placebo
  Interventions: Drug: FGI-101-1A6

INTERVENTIONS:
Drug: FGI-101-1A6 — anti-TSG101 human monoclonal antibody, single dose

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the anti-TSG101 human monoclonal antibody (FGI-101-1A6)when administered intravenously to healthy volunteers.

DETAILED DESCRIPTION:
Primary -

- To compare the safety profile of a single intravenous administration of FGI-101-1A6 as compared with Placebo

Secondary

* To evaluate the pharmacokinetics (PK) of a singel intravenous administration of FGI-101-1A6
* To evaluate the immunogenicity of FGI-101-1A6

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ages 18-45
* Normal laboratory (blood tests) results

Exclusion Criteria:

* Prior immunization with live-attenuated vaccines

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Safety assessments | 60 days following infusion
  Safety will be assessed by collecting data (physical exams, adverse event reporting, lab testing/analysis) and concomitant medications at each visit from pre-infusion period through post-infusion day 60, or the early withdrawal, if applicable

SECONDARY OUTCOMES:
Pharmacokinetic analysis (PK) | 60 days following infusion
  PK parameters will be determined for a single administration of FGI-101-1A6 as measured by an immunoassay for FGI-101-1A6
Immunogenicity | From day 1 up to day 60 following infusion
  Immunogenicity will be measured by testing serum on anti-FGI-101-1A6 generation

CONTACTS AND LOCATIONS:
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States